CLINICAL TRIAL: NCT01585597
Title: Phase 1 Study of Mild Induced Hypothermia After Endovascular Revascularization in Acute Ischemic Stroke of the Anterior Circulation
Brief Title: Reperfusion With Cooling in Cerebral Acute Ischemia
Acronym: ReCCLAIM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Christopher M. Horn, MD, Assistant Professor of Neurology and Neurosurgery, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00056889; MSNC 01 (Other: Other)
Record Dates: First submitted 2012-04-22; First posted 2012-04-26 (Estimated); Results first posted 2014-08-01 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Stroke, Acute
Keywords: Ischemic Stoke; Endovascular Reperfusion; Reperfusion Injury; Mild hypothermia
MeSH Terms: conditions — Stroke; Reperfusion Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mild Hypothermia (Experimental): Reduction of body temperature to 34 degrees centigrade. This will be accomplished using the Zoll Coolguard .
  Interventions: Device: Zoll- Coolgaurd 3000

INTERVENTIONS:
Device: Zoll- Coolgaurd 3000 — Goal temperature of 33 degrees Centigrade for a duration of 12 hours and then actively rewarmed by 0.2 degrees Centigrade per hour.

SUMMARY:
The purpose of this study is to determine whether reducing a patients body temperature (mild hypothermia of 33 degrees Centigrade) will significantly reduce the risk of brain injury (notably reperfusion injury and hemorrhagic conversion) in patients that have suffered a significant interruption of blood flow to an area of brain (occlusion of large proximal cerebral artery) and have undergone successful removal of that interruption (revascularization).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85 years old
* Symptoms consistent with an ischemic stroke with a large vessel occlusion (MCA, ICA-terminus) as determined by vascular imaging
* ASPECTS score of 5-7 on non-contrast CT of the brain
* Ability to undergo endovascular reperfusion therapy
* Must have no contraindications to general anesthesia
* A pre-treatment modified Rankin Score of 0 or 1
* Arterial puncture performed under 8 hours from symptom onset or last seen normal
* Immediate post reperfusion CT scan shows no hemorrhage

Exclusion Criteria:

* Bleeding diathesis with a platelet count < 50,000 or INR > 1.5
* Involved in another clinical trial
* History of dementia
* End stage renal disease on hemodialysis
* History of ventricular dysrhythmias
* Life threatening medical condition precluding survival under 6 months
* Presence of an IVC filter
* Contrast dye allergy with history of anaphylaxis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rishi Gupta, MD, Study Director — Emory University
Locations (1):
- Marcus Stroke and Neuroscience Center at Grady Memorial Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Horn CM, Sun CH, Nogueira RG, Patel VN, Krishnan A, Glenn BA, Belagaje SR, Thomas TT, Anderson AM, Frankel MR, Schindler KM, Gupta R. Endovascular Reperfusion and Cooling in Cerebral Acute Ischemia (ReCCLAIM I). J Neurointerv Surg. 2014 Mar;6(2):91-5. doi: 10.1136/neurintsurg-2013-010656. Epub 2013 Mar 6. PMID 23468538

RESULTS

PARTICIPANT FLOW:
Groups:
- Mild Hypothermia: Reduction of body temperature to 34 degrees centigrade.
  Zoll- Coolgaurd 3000: Goal temperature of 33 degrees Centigrade for a duration of 12 hours and then actively rewarmed by 0.2 degrees Centigrade per hour.
Period: Overall Study
Arm/Group | Mild Hypothermia
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Mild Hypothermia
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Reperfusion Injury \ Hemorrhagic Transformation
Description: Asymptomatic and symptomatic Hemorrhages defined as homogenous density occupying >30% of the infarct zone with mass effect
Time Frame: 24 Hours
Measure: Number; unit: participants
Arm/Group | Mild Hypothermia
Number analyzed (Participants) | 20
participants | 3

2. Secondary Outcome: Modified Rankin Scale 0-2
Description: Modified Rankin Score 0=no symptoms
  1. no significant disability
  2. slight disability needs help
  3. moderate disability
  4. moderate serve disability
  5. severe disability 0-2 = good outcome 3-5= poor outcome
Time Frame: 90 days post hospitalization
Measure: Number; unit: participants Modified Rankin Scal 0-2
Arm/Group | Mild Hypothermia
Number analyzed (Participants) | 20
participants Modified Rankin Scal 0-2 | 20

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Mild Hypothermia
Serious Adverse Events (participants affected / at risk) | 8/20
Other Adverse Events (participants affected / at risk) | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mild Hypothermia (N=20)
Pneumonia (Infections and infestations) | 5 (5)
Bacteremia (Infections and infestations) | 1 (1)
Deep Venous Thrombosis (Blood and lymphatic system disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No